CLINICAL TRIAL: NCT04134624
Title: EMS Prehospital Blood Culture Collection and Antibiotic Administration: A Two-Phase Pilot Project to Reduce Mortality in Patients With Severe Sepsis and Septic Shock
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment for this study was halted in February 2020 due to the COVID-19 pandemic. The study team was unable to continue enrollment due to decreased volumes (and the fact that COVID-19 mimics some of the signs and symptoms of severe sepsis)
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A19-118
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2019-10

CONDITIONS: Sepsis; Sepsis, Severe; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: This is a stepwise study with two phases. In phase 1, all eligible patients have a blood culture collected. In phase 2, eligible patients have a blood culture collected and antibiotics started in the prehospital setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehospital intervention (Active Comparator): All subjects enrolled in this study will receive a sepsis intervention bundle in the prehospital setting, including blood cultures, IV fluids, and antibiotics. These patients will be compared to historical controls.
  Interventions: Other: Sepsis care bundle
- Control arm (No Intervention): Historical controls without prehospital sepsis intervention.

INTERVENTIONS:
Other: Sepsis care bundle — Initiation of sepsis care bundle in prehospital setting, including collection of blood cultures, administration of antibiotics, and initiation of IV fluids
  Arms: Prehospital intervention

SUMMARY:
This study is designed to improve the outcomes for patients suffering from severe sepsis and septic shock (SS/SS) by decreasing the time from first medical contact to antibiotic administration. This is a stepwise study that aims to demonstrate the ability of paramedics to accurately obtain blood cultures prior to hospital arrival, administer a broad spectrum antibiotic and initiate IV fluid resuscitation in patients meeting predefined criteria for SS/SS.

DETAILED DESCRIPTION:
This study is designed to improve the outcomes for patients suffering from severe sepsis and septic shock (SS/SS) by decreasing the time from first medical contact to antibiotic administration. This is a pilot project. This is a stepwise study that will build on previously published literature to demonstrate the ability of paramedics to accurately obtain blood cultures prior to hospital arrival, administer a broad spectrum antibiotic and initiate IV fluid resuscitation in patients meeting predefined criteria for SS/SS. The primary aim is to take processes that have been developed for use in this patient population during Emergency Department care and to advance these same processes "downrange" to initiate them prior to hospital arrival. Early antibiotic administration has been shown to decrease mortality in a time dependent fashion when implemented in hospitalized patients. The investigators hypothesize that initiating antibiotics prior to hospital arrival will improve morbidity and mortality while also addressing quality metrics that are publicly reported for this patient population.

This pilot study will be conducted in two consecutive phases, responding to the following aims.

Aim 1: Evaluate the feasibility that paramedics can obtain blood cultures from general patients prior to hospital arrival with a contamination rate that is statistically equivalent to that for blood cultures obtained in Emergency Department.

Aim 2 (primary aim): Investigate whether prehospital paramedic initiated broad spectrum antibiotics, administered after blood cultures are obtained, will result in improved mortality rates for patients, when compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (blood culture contamination rate quantification phase)

1. Hemodynamically stable patients ≥18 years old being transported by Lakeview EMS to Lakeview Hospital who will have an intravenous access established as part of their routine prehospital care are eligible for this study.
2. English speaker

Phase 2 (blood cultures + antibiotics prehospital)

a. Patients with fever >38oC + ≥2 qSOFA who are being transported to Lakeview Hospital that originate as a 911 call

Exclusion Criteria:

Phase 1:

1. Patients age <18 years
2. Hemodynamic instability
3. Prisoners

Phase 2:

1. Documented allergy to Penicillin or inability to determine patient's medication allergies
2. Prisoners
3. Pregnant patients
4. Patients being transferred from one hospital to another
5. Non-English speakers

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
In hospital mortality | Through duration of hospitalization, average 1 week
  Mortality during hospital admission following enrollment
ICU length of stay | Through duration of ICU stay, average 3 days
  Length of stay in ICU during hospital admission following enrollment
Hospital length of stay | Through duration of hospitalization, average 1 week
  Length of stay of hospitalization following enrollment
30 day mortality | 30 days
  Mortality 30 days following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Burnett, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Lakeview Hospital, Stillwater, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kadri SS, Rhee C, Strich JR, Morales MK, Hohmann S, Menchaca J, Suffredini AF, Danner RL, Klompas M. Estimating Ten-Year Trends in Septic Shock Incidence and Mortality in United States Academic Medical Centers Using Clinical Data. Chest. 2017 Feb;151(2):278-285. doi: 10.1016/j.chest.2016.07.010. Epub 2016 Jul 22. PMID 27452768
- [Background] Howell MD, Davis AM. Management of Sepsis and Septic Shock. JAMA. 2017 Feb 28;317(8):847-848. doi: 10.1001/jama.2017.0131. No abstract available. PMID 28114603
- [Background] Kumar A, Haery C, Paladugu B, Kumar A, Symeoneides S, Taiberg L, Osman J, Trenholme G, Opal SM, Goldfarb R, Parrillo JE. The duration of hypotension before the initiation of antibiotic treatment is a critical determinant of survival in a murine model of Escherichia coli septic shock: association with serum lactate and inflammatory cytokine levels. J Infect Dis. 2006 Jan 15;193(2):251-8. doi: 10.1086/498909. Epub 2005 Dec 13. PMID 16362889
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- [Background] Liu VX, Fielding-Singh V, Greene JD, Baker JM, Iwashyna TJ, Bhattacharya J, Escobar GJ. The Timing of Early Antibiotics and Hospital Mortality in Sepsis. Am J Respir Crit Care Med. 2017 Oct 1;196(7):856-863. doi: 10.1164/rccm.201609-1848OC. PMID 28345952
- [Background] Gaieski DF, Mikkelsen ME, Band RA, Pines JM, Massone R, Furia FF, Shofer FS, Goyal M. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53. doi: 10.1097/CCM.0b013e3181cc4824. PMID 20048677
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] Peake SL, Delaney A, Bellomo R; ARISE Investigators. Goal-directed resuscitation in septic shock. N Engl J Med. 2015 Jan 8;372(2):190-1. doi: 10.1056/NEJMc1413936. No abstract available. PMID 25564906
- [Background] Lane D, Ichelson RI, Drennan IR, Scales DC. Prehospital management and identification of sepsis by emergency medical services: a systematic review. Emerg Med J. 2016 Jun;33(6):408-13. doi: 10.1136/emermed-2015-205261. Epub 2016 Feb 10. PMID 26864327
- [Background] Walchok JG, Pirrallo RG, Furmanek D, Lutz M, Shope C, Giles B, Gue G, Dix A. Paramedic-Initiated CMS Sepsis Core Measure Bundle Prior to Hospital Arrival: A Stepwise Approach. Prehosp Emerg Care. 2017 May-Jun;21(3):291-300. doi: 10.1080/10903127.2016.1254694. Epub 2016 Dec 5. PMID 27918869